CLINICAL TRIAL: NCT02021084
Title: The Effect of Probiotics on Response to Therapy and on Adverse Effect in Patients Treated With Colchicine for Familial Mediterranean Fever.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient enroled
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, yonatan butbul MD, Butbul Aviel Yonatan, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0173-13-RMB CTIL
Record Dates: First submitted 2013-10-29; First posted 2013-12-27 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Familial Mediterranean Fever (FMF )
Keywords: Familial Mediterranean Fever (FMF), probiotics
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo, response, adverse effect (Placebo Comparator): children (5-17 years old) with FMF that are currently followed in the pediatric rheumatology clinic at Mayer children hospital Israel Haifa that are being treated with colchicine and suffering from either gastrointestinal adverse effect or partial response to colchicine.in the first 3 month patients will be followed with no interventions and will be required to record all there FMF episodes and their GIT adverse effect, in the second period the patients will be randomly divided into two groups patients that will received placebo arm one and patients that will receive probiotics arm two.
  Interventions: Dietary Supplement: Placebo
- probiotic, response, adverse effect (Active Comparator): children (5-17 years old) with FMF that are currently followed in the pediatric rheumatology clinic at Mayer children hospital Israel Haifa that are being treated with colchicine and suffering from either gastrointestinal adverse effect or partial response to colchicine.in the first 3 month patients will be followed with no interventions and will be required to record all there FMF episodes and their GIT adverse effect, in the second period the patients will be randomly divided into two groups patients that will received placebo arm one and patients that will receive probiotics arm two.
  Interventions: Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: probiotic — Probiotics group - patients will received probiotics Bio -25 including 11 types of bacteria total of 25 billion germs in each capsule, patients will received one capsule a day for 3 month.
  Other Names: Bio 25
  Arms: probiotic, response, adverse effect
Dietary Supplement: Placebo — Placebo group - patients will received placebo patients will received one capsule a day for 3 month.
  Arms: placebo, response, adverse effect

SUMMARY:
Colchicine is the drug of choice to treat patients with Familial Mediterranean Fever (FMF ), some of the patients treated with colchicine may suffer from gastrointestinal (GIT) adverse effect such as diarrhea and abdominal pain especially in the higher dose.

5-10% of the patients with FMF that have been treated with colchicine may have partial or no response to this therapy.

Aim of our study: the aim of our study is :.1to evaluate the efficacy of probiotics in reducing the number of adverse effect in patients with FMF that are being treated with colchicine and suffering from GIT adverse effect.

.2 To evaluate the efficacy of probiotics in reducing the number of FMF attacks in children with FMF that has been treated with colchicine with only partial response.

Methods: the study will be done among children (5-17 years old) with FMF that are currently followed in the pediatric rheumatology clinic at Mayer children hospital Israel Haifa that are being treated with colchicine and suffering from either GIT adverse effect or partial response to colchicine.

The study is design to be double blind placebo control, in the first 3 month patients will be with no therapy and will be required to record all there FMF episodes and their GIT adverse effect, in the second period the patients will be randomly divided into two groups 1.patients that will received placebo (group 1) and the 2. Probiotics group - patients will received probiotics (Bio -25 including 11 types of bacteria L.acidophilus, B.bifidum , L.rhamnosus, L.lactis, L.casei, B.breve, B.thermophilus, B.longum, L.paracseis, L.plantarum, B.infantis), both for three month, during this period patient will be required to record their gastrointestinal symptoms and other symptoms that may be related to FMF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of FMF
* Age 5-18 years
* Colchicine therapy
* Gastrointestinal adverse effect or recurrent FMF attacks on colchicine

Exclusion Criteria:

• Severe immune deficiency

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The number of gastrointestinal adverse effect related to colchicine therapy after adding probiotics to colchicine therapy. | 6 months after enrollment assumed to be at 12/2014
  The number of gastrointestinal adverse effect will be measured 3 months before starting the intervention and after 3 months patients will received either placebo or probiotics the measures will be :
  1. Number of days with at least one episode of loose stool.
  2. Number of days with abdominal pain not related to FMF attacks.

SECONDARY OUTCOMES:
Number of FMF attacks after adding the probiotics to the colchicine therapy | 6 months after enrollment assumed to be at 12/2014
  The number of attacks will be measured 3 months before starting the intervention and after 3 months patients will received either placebo or probiotics .
  Attacks will defined as fever with one of the above : a. abdominal pain b.pleuritic chest pain c.arthritis d.erysipelas like .

CONTACTS AND LOCATIONS:
Overall Officials: Butbul Yonatan, M.D, Principal Investigator — Rambam medical center, Mayers childrens hospital